CLINICAL TRIAL: NCT03903861
Title: Galactose Mediated Glycogen Resynthesis and the Effects on Metabolism During Subsequent Exercise
Brief Title: Galactose Mediated Glycogen Resynthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ERN_19-0308
Record Dates: First submitted 2019-03-29; First posted 2019-04-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity | interventions — Glucose; Galactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glucose alone (Experimental): Participants will complete a glycogen depleting bout of exercise followed by the provision of glucose-alone over 4 hours of recovery before a subsequent bout of exercise.
  Interventions: Other: Glucose alone
- Galactose alone (Experimental): Participants will complete a glycogen depleting bout of exercise followed by the provision of galactose-alone over 4 hours of recovery before a subsequent bout of exercise.
  Interventions: Other: Galactose alone
- Glucose and galactose (Experimental): Participants will complete a glycogen depleting bout of exercise followed by the provision of glucose and galactose over 4 hours of recovery before a subsequent bout of exercise.
  Interventions: Other: Glucose and galactose

INTERVENTIONS:
Other: Glucose alone — Young men or women will complete a glycogen depleting bout of exercise followed by the provision of glucose-alone over 4 hours of recovery before a subsequent bout of exercise.
  Arms: Glucose alone
Other: Galactose alone — Young men or women will complete a glycogen depleting bout of exercise followed by the provision of galactose-alone over 4 hours of recovery before a subsequent bout of exercise.
  Arms: Galactose alone
Other: Glucose and galactose — Young men or women will complete a glycogen depleting bout of exercise followed by the provision of glucose and galactose over 4 hours of recovery before a subsequent bout of exercise.
  Arms: Glucose and galactose

SUMMARY:
This study will compare short-term post-exercise muscle glycogen synthesis following combined galactose-glucose, glucose alone or galactose alone ingestion.

DETAILED DESCRIPTION:
Lactose, the sugar contained within milk, consists of glucose and galactose. Post-exercise consumption of a carbohydrate mixture containing glucose with galactose has been shown to accelerate liver glycogen repletion as compared to glucose-only provision. However, the extent to which galactose-glucose combinations influence post-exercise muscle glycogen storage has yet to be determined.

Therefore, this study will investigate whether short-term muscle glycogen storage after strenuous endurance exercise is enhanced by combined galactose-glucose or glucose only ingestion as compared to the ingestion of galactose alone.

ELIGIBILITY:
Inclusion Criteria:.

* Body mass index in the range: 18.5 - 27.5 kg/m2
* Participates in endurance-based exercise (e.g. cycling, running, rowing) at least 3 times per week
* Aerobic fitness: VO2max >45 ml/kg/min (men), >40 ml/kg/min (women)

Exclusion Criteria:

* Lidocaine allergy
* Current participation in another scientific/clinical study
* Bleeding disorder/s
* Current or recent smoker to include vaping (last 60 days)
* Vegan
* Existence of food intolerances
* Poor recent health as indicated in the general health questionnaire
* Engage in uncommon eating practices (e.g. sustained periods of fasting)
* Diagnosed with galactosemia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Muscle glycogen synthesis rates (mmol/kg/dm/h) | 4 hours
  Muscle glycogen synthesis rates over the post-exercise recovery period

SECONDARY OUTCOMES:
Carbohydrate oxidation rates (g/min) | Up to 90 minutes
  Total, exogenous and endogenous carbohydrate oxidation during a secondary bout of exercise
Fat oxidation rates (g/min) | Up to 90 minutes
  Fat oxidation during a secondary bout of exercise
Plasma glucose (mmol/L) | Up to 6 hours
  Plasma glucose during the post-exercise recovery period and during a secondary bout of exercise
Serum insulin (mU/L) | Up to 6 hours
  Serum insulin during the post-exercise recovery period and during a secondary bout of exercise
Plasma galactose (mmol/L) | Up to 6 hours
  Plasma galactose during the post-exercise recovery period and during a secondary bout of exercise
Plasma lactate (mmol/L) | Up to 6 hours
  Plasma lactate during the post-exercise recovery period and during a secondary bout of exercise
Plasma non-esterified fatty acids (mmol/L) | Up to 6 hours
  Plasma non-esterified fatty acids during the post-exercise recovery period and during a secondary bout of exercise
Plasma glycerol (umol/L) | Up to 6 hours
  Plasma glycerol during the post-exercise recovery period and during a secondary bout of exercise
Plasma glucagon (pmol/L) | Up to 6 hours
  Plasma glucagon during the post-exercise recovery period and during a secondary bout of exercise

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Wallis, PhD, Principal Investigator — University of Birmingham
Locations (1):
- School of Sport, Exercise and Rehabilitation Sciences, Birmingham, West Midlands, United Kingdom